CLINICAL TRIAL: NCT05876286
Title: Sleep and Memory Consolidation in Adults With Attention Deficit Hyperactivity.
Acronym: HYPNOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/22/0488
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Sleep; Memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Deficit Disorder With Hyperactivity (Experimental): Patients with Attention Deficit Disorder With Hyperactivity. Same examinations than control group
  Interventions: Other: Neurological examinations
- Control (Active Comparator): Healthy volunteers Same examinations than Attention Deficit Disorder With Hyperactivity group
  Interventions: Other: Neurological examinations

INTERVENTIONS:
Other: Neurological examinations — Neurological, neuropsychological, polysomnography examinations and multiple sleep latency test. The protocol is divided into three visits.

SUMMARY:
Attention Deficit Disorder With Hyperactivity is associated with deficits in cognition and sleep. In healthy adults, memory consolidation processes are related to sleep spindle activity in the sleep electroencephalogram. This association is poorly characterized in adults with attention deficit hyperactivity. In this study, the purpose is to characterize sleep microarchitecture disorders through the analysis of different stage of sleep EEG activity during a polysomnographic examination in adult with mixed Attention Deficit Disorder With Hyperactivity presentation compared to healthy.

ELIGIBILITY:
Inclusion Criteria for all participants:

* Age from 18 to 45 years old
* Affiliated to the French health care system

Inclusion Criteria for attention deficit hyperactivity disorder patients:

* meeting Diagnostic and Statistical Manual (DSM)-5 criteria for mixed attention deficit hyperactivity disorder presentation without drug treatment for attention deficit hyperactivity disorder.

Exclusion Criteria for all participant:

* People not able to give consent, neurological disease (other than neurodevelopmental disorders; or any other serious disease (cancer, addiction, systemic disease)), untreated sleep apnea, major depression (Beck inventory > 15), untreated restless leg syndrome; pregnancy in progress or wish to become pregnant during the study or breastfeeding woman, drug treatment including benzodiazepine, neuroleptic or antidepressant before inclusion.

Exclusion Criteria for healthy volunteers:

* Subjective cognitive and/or sleep complaint.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference in signal power (db or μV 2) in the sigma frequency bands in N2 sleep | 1 day
  difference between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie PLANTON, PhD, Principal Investigator — University Hospital, Toulouse